CLINICAL TRIAL: NCT02388074
Title: Sputum Labeling Utilizing Synthetic Meso Tetra (4-Carboxyphenyl) Porphine (TCPP) for Detection of Lung Cancer
Brief Title: Sputum Labeling Utilizing Synthetic Meso-Tetra (4-Carboxyphenyl) Porphine (TCPP) for Detection of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bioAffinity Technologies Inc. (Industry)
Collaborators: Radiology Associates of Albuquerque (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MODA-002
Record Dates: First submitted 2015-03-04; First posted 2015-03-13 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Porphyrin; Fluorescence; Diagnostic; Sputum Cytology; Early Detection
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyPath® Assay of Deep-Lung Sputum Sample (Experimental): Deep-lung sputum was obtained from healthy individuals who had no known lung disease, was labeled with TCPP and evaluated to detect red fluorescent [ie, cancer] cells (RFCs) from deep-lung sputum samples.
  Interventions: Device: CyPath®

INTERVENTIONS:
Device: CyPath® — CyPath® diagnostic assay for the early detection of lung cancer using sputum

SUMMARY:
This is a single center study to assess the efficacy of CyPath® Early Detection Lung Cancer Assay to detect lung cancer cells from deep lung sputum.

DETAILED DESCRIPTION:
Meso Tetra (4-Carboxyphenyl) Porphine (TCPP) is a porphyrin that can label cancer cells by reacting to the increased number of low-density lipoproteins coating the surface of cancer cells and the porous nature of the cancer cell membrane, causing the cell to fluoresce under specific wavelengths of light. The primary objective of this clinical trial is to determine the the presence or absence of red fluorescent [ie, cancer] cells (RFCs) from deep-lung sputum samples using the CyPath® Early Lung Cancer Detection Assay from one cohort of Participants who are healthy. The results from this trial will be compared with two additional cohorts of Participants including individuals at high risk for lung cancer and individuals diagnosed with lung cancer. Collection of the sputum samples from high-risk individuals and lung cancer patients is complete (NCT00894127).

Participants who satisfy the inclusion/exclusion criteria will be enrolled into the study and assigned to the healthy cohort. The sputum samples will be collected at the study site or at the Participant's home after explanation of the collection procedure by study staff. Samples will be identified with an identification number blinding the sample identity. Each subject's sputum specimen will be processed onto 13 microscope slides at the University of Texas Health Science Center of San Antonio (UTHSCSA) Laboratory. The UTHSCSA laboratory will process each sputum sample onto slides using the ThinPrep T2000 processor for use in the CyPath® Early Lung Cancer Detection Assay.

Twelve slides from each sputum sample will be labeled with CyPath®. One slide will be used to preform PAP staining for the presence of macrophages. Macrophages are an indication that the sputum sample is from deep within the lungs. A cytopathologist will review the slide and record results on a specimen adequacy form. bioAffinity researchers who will be blinded as to the Participant's identity will perform the CyPath® labeling and scoring of the slides. The study results of the healthy cohort will be used for comparison with the results of a closed study in which the sputum from individuals at high risk of lung cancer and individuals diagnosed with lung cancer was compared.

Findings of the CyPath® assay will not be used in the diagnosis or treatment of Participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have never smoked nor have known lung diseases

Exclusion Criteria:

* Severe obstructive lung disease
* Angina with minimal exertion
* Pregnancy
* Have or have had cancer other than lung cancer
* Worked in the mining Industry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Patriquin, MD, Principal Investigator — Radiology Associates of Albuquerque
Locations (1):
- Radiology Associates of Albuquerque (RAA), Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at Radiology Associates of Albuquerque (RAA), New Mexico during the recruitment period of March 2015 to April 20, 2015
Groups:
- CyPath® Assay of Deep-Lung Sputum Sample: Deep-lung sputum was obtained from healthy individuals who had no known lung disease, was labeled with TCPP and evaluated to detect red fluorescent [i.e., cancer] cells (RFCs) from deep-lung sputum samples.
  CyPath®: CyPath® diagnostic assay for the early detection of lung cancer using sputum
Period: Overall Study
Arm/Group | CyPath® Assay of Deep-Lung Sputum Sample
Started | 25
Completed | 22
Not Completed | 3
Not completed — Lost in Transit | 2
Not completed — Sample Not Returned | 1

BASELINE CHARACTERISTICS:
Arm/Group | CyPath® Assay of Deep-Lung Sputum Sample
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Red Fluorescent [i.e., Cancer] Cells (RFCs) in Sputum From Healthy Participants
Description: The presence or absence of red fluorescent (RFCs) cancer cells was evaluated in sputum samples from healthy individuals labeled with CyPath®.
  Testing for the study was performed at one study center to collect sputum samples from healthy individuals who have no known lung disease. Comparison of sputum specimens from one cohort of Participants who are healthy with two additional cohorts of Participants, including individuals at high risk for lung cancer and individuals diagnosed with lung cancer, that has already been completed.
Time Frame: 2 months
Population: 22 participants were evaluated by a cytopathologist. Of these 22, PAP-stained slides of 3 participants were unreadable, 14 participants had provided samples that were confirmed by PAP as inadequate and only 5 slides were confirmed by PAP as adequate deep lung sputum samples. These 5 samples were evaluated for the presence of RFCs.
Measure: Mean (Standard Deviation); unit: number of RFCs per participant
Arm/Group | CyPath® Assay of Deep-Lung Sputum Sample
Number analyzed (Participants) | 5
number of RFCs per participant | 0 (0)

ADVERSE EVENTS:
Arm/Group | CyPath® Assay of Deep-Lung Sputum Sample
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No